CLINICAL TRIAL: NCT04027738
Title: Efficacy of a Single Intraarticular Injection of Platelet-Rich Plasma for the Treatment of Early Knee Osteoarthritis
Brief Title: a Single Intraarticular Injection of PRP for Early Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, Director of Neutorehabilitation, MD,Department of Physical Medicine and Rehabilitation, Kaohsiung Veterans General Hospital, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS106-131
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee; Osteoarthritis; Platelet rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection (Experimental): The patients received a single 3-ml injection of PRP.
  Interventions: Other: PRP

INTERVENTIONS:
Other: PRP — The patients received a single 3-ml injection of PRP. Approximately 10-mL of venous blood was drawn from each patient and centrifuged using an Arthrex autologous conditioned plasma (ACP) kit (a low-leukocyte ACP system), spun at a speed of 1500 rpm for 5 minutes. The platelet concentration obtained was approximately 2-3 times greater than the baseline platelet concentration.

SUMMARY:
This study aimed to investigate the efficacy of a single intraarticular injection of PRP for the treatment of early knee OA.

DETAILED DESCRIPTION:
Platelet-rich plasma (PRP) has been reported to be effective for the treatment of knee osteoarthritis (OA). This study aimed to investigate the efficacy of a single intraarticular injection of PRP for the treatment of early knee OA.

In a prospective trial with 6-month follow-up, patients with early knee OA were recruited and received a single intraarticular PRP injection. Several outcomes were measured.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-70 years
* symptomatic knee OA with pain for at least 6 months despite conservative treatment such as analgesics, NSAIDs and/or physical therapy
* average knee pain of at least 30 mm on a 100-mm visual analog (VAS) scale
* grade 1 or 2 knee OA according to the Kellgren-Lawrence grading system based on -radiographs taken within the previous 6 months
* Radiological evidence of bilateral knee OA was accepted if global pain VAS in the contralateral knee was less than 30 mm.

Exclusion Criteria:

* previous orthopedic surgery on the spine or lower limbs
* disabling OA of either hip or foot
* knee instability or marked valgus/varus deformity
* history of severe knee trauma; intraarticular injections into the knee in the past 6 months
* infections or skin diseases around the target knee
* women ascertained or suspected pregnancy or lactating
* presence of malignancy, hematological disease, collagen vascular diseases, or autoimmune diseases;
* therapy with anticoagulants or anti-aggregating agent
* serious medical conditions that would interfere with the assessments during the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
VAS pain | 6 months
  The primary outcome was the change from baseline in the VAS pain score at 6 months. The patient rated the average severity of knee pain on knee movement over the previous week on a 0-100 mm VAS (0=no pain to 100=worst possible pain)

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC, Likert Scale) is a 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function [17]. The patient answers the questions and then receives a cumulative score in each of the 3 areas (pain, 0-20; stiffness, 0-8; physical function, 0-68). Total score is 96 and higher scores indicate worse outcomes.
Lequesne index | 6 months
  Lequesne index is used to assess severity of knee symptoms during the last week .It is validated and includes the measurement of pain (5 items), walking distance (2 items), and activities of daily living (4 items). Maximal score is 24 and higher scores represent worse function.
Single-leg stance test (SLS) | 6 months
  Single-leg stance test (SLS) is done by raising one foot up without touching it to the supported lower extremity with target knee and maintain balance for as long as possible. Each participant performed 3 trials, and the best result of the 3 trials was recorded
Patients satisfaction | 6 months
  Patients were asked to rate their treatment satisfaction compared to the preinjection condition, using a 100 mm VAS (0= completely dissatisfied, 100=completely satisfied)
safety assessment | during the study, for 6 months
  The safety assessment was based on adverse events reported by the patients during the study and physical findings by the evaluator at each follow-up. The occurrence of adverse events was recorded, including duration, action taken and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Fen Sun, MD, Principal Investigator — Kaohsiung Veterans General Hospital, Taiwan
Locations (1):
- Department of Physical Medicine and Rehabilitation, Veterans General Hospital,, Kaohsiung City, Taiwan